CLINICAL TRIAL: NCT05016765
Title: Open Trial of Median Nerve Stimulation for Treatment of Tourette Syndrome
Brief Title: Open-label MNS for Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Kevin J. Black, M.D., Principal Investigator, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Open-label MNS; UL1TR002345 (NIH)
Record Dates: First submitted 2021-08-09; First posted 2021-08-23 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Tourette Syndrome; Tic Disorder, Chronic Motor or Vocal
Keywords: Tourette; tic; Transcutaneous Electric Nerve Stimulation; Median Nerve
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Tics

STUDY DESIGN:
Intervention Model Description: All participants will receive MNS at 12 Hz, pulse width 200µs. After initial threshold determination and training on device usage, individual participants will choose duration and intensity of treatment depending on their momentary symptom severity and history of response to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active MNS (Experimental): Active, self-directed electrical stimulation of the right median nerve
  Interventions: Device: Active, self-directed electrical stimulation of the median nerve

INTERVENTIONS:
Device: Active, self-directed electrical stimulation of the median nerve — Electrical stimulation of the median nerve (12 Hz, pulse width 200µs), initially at the threshold needed to see movement of the right thumb with stimulation. After initial training with the device and education in the rationale for suprathreshold stimulation, participants will choose timing and intensity of stimulation based on their momentary symptom severity and their experience with the treatment since the beginning of the study. Participant can choose right or left median nerve (we will suggest their nondominant hand to minimize interference with daily activities).
  Other Names: Rhythmic MNS

SUMMARY:
A recent report (Morera Maiquez et al 2020) described reduced tic severity in people with Tourette syndrome during 1-minute epochs of median nerve stimulation (MNS) at 10 Hz. Among the various questions still to be answered is the question of whether a device to administer MNS is practical for use in a chronic, real-world setting. This study will recruit participants who complete the clinic-based, blinded, randomized controlled trial, https://clinicaltrials.gov/ct2/show/NCT04731714, to determine the real-world usage and apparent utility of median nerve stimulation in people with chronic tics.

DETAILED DESCRIPTION:
Chronic tic disorders (CTD), including Tourette syndrome (TS), are associated with a substantially reduced quality of life (Evans et al 2016). Medication treatments are no more than 50-60% effective in randomized, controlled trials (RCTs), and are often discontinued due to unacceptable side effects (Thomas and Cavanna 2013). Behavioral therapies require ability to participate in therapy and a specially trained therapist (Scahill et al 2013), but weekly visits to psychologists are impractical for many Americans, especially in rural areas (Lin et al 2016). Patients strongly desire new treatment options (Cuenca et al 2015).

In June, 2020, Stephen Jackson's group at the University of Nottingham published a fascinating report in Current Biology on a potential novel treatment for tics (Morera Maiquez et al 2020). The radical new idea arose from observations associating movement inhibition with 8-14 Hz activity in motor cortex. They first showed that rhythmic 12 Hz peripheral stimulation of the median nerve evoked synchronous contralateral EEG activity over primary sensorimotor cortex, whereas arrhythmic stimulation at the same mean rate did not. As hypothesized, median nerve stimulation (MNS) at 12 Hz created small but statistically significant effects on initiation of voluntary movements. Importantly, they also demonstrated that this stimulation did not meaningfully impair concentration, suggesting that the effect did not operate through simple distraction. They went on to test 10 Hz MNS in 19 TS patients, and demonstrated using blinded video ratings a significant reduction in tic number and severity during 1-minute stimulation epochs vs 1-minute no-stimulation epochs. They noted that in some participants, benefit lasted beyond the end of the stimulation epoch [personal correspondence]. Videos accompanying the publication showed dramatic benefit during MNS in some subjects. Although the authors appropriately noted the steps needed to generalize these results to clinical practice, news reports already have led a number of TS patients to contact them asking for treatment. The Nottingham group has referred such inquiries from the U.S. to me as leader of our Wash.U. Tourette Association of America (TAA) Center of Excellence.

Among the various questions still to be answered is the question of whether such a device would be practical for use in the real world. This study will supply participants with a commercially available transcutaneous electrical nerve stimulation (TENS) units to use for median nerve stimulation as described in the Nottingham study. Participants will be told to use the device as much or as little as desired to see how such stimulation might be utilized in the real world.

Here the investigators propose (a) to determine the real-world usage and apparent utility of stimulation in people with chronic tics, and (b) to determine momentary self-rated efficacy and side effects of stimulation. The investigators will also compare results from this study to those from the "Peripheral induction of inhibitory brain circuits to treat Tourette's: pilot" study, from which participants will be drawn, in order to compare laboratory and real-world efficacy.

Aim 1. Determine the real-world usage and apparent utility of stimulation in people with chronic tics. Participants will be allowed to choose when and for how long to use the stimulation, thus simulating how patients would use the stimulation in their daily lives.

Aim 2. Determine momentary self-rated efficacy and side effects of stimulation, using surveys taken at the beginning and end of stimulation periods, as well as twice daily when prompted.

Aim 3. Compare results of this trial with those from "Peripheral induction of inhibitory brain circuits to treat Tourette's: pilot." Participants in this study will have been drawn from completers of the "peripheral induction" blinded RCT, allowing for clear comparisons between the laboratory conditions of the first study and the real-world conditions of the second.

Completion of these Aims will provide practical information that can inform a future, controlled clinical trial of chronic MNS delivered by a portable device.

ELIGIBILITY:
Inclusion Criteria:

* Completed participation in the study called "Peripheral induction of inhibitory brain circuits to treat Tourette's: pilot"
* Informed consent by adult participant, or assent by child and informed consent by guardian

Exclusion Criteria:

* Has an implanted device that could be affected by electrical current
* Pregnancy known to participant or (for children) to the parent
* Severe or unstable systemic illness
* Factors (such as exaggerated symptom report) that in the judgment of the principal investigator may make the outcome measures inaccurate
* Judged by investigator to be unlikely to complete study procedures

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Black, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, Movement Disorders Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD other than PHI (protected health information) will be shared on OSF.io or as a supplement to publication of results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available within 6 months after publication of key results
Access Criteria: Individual participant data (IPD) will be freely available under a CC0 license (Creative Commons public domain dedication, https://creativecommons.org/publicdomain/zero/1.0/).
URL: https://osf.io/2y7fs/

REFERENCES:
- [Background] Evans J, Seri S, Cavanna AE. The effects of Gilles de la Tourette syndrome and other chronic tic disorders on quality of life across the lifespan: a systematic review. Eur Child Adolesc Psychiatry. 2016 Sep;25(9):939-48. doi: 10.1007/s00787-016-0823-8. Epub 2016 Feb 15. PMID 26880181
- [Background] Thomas R, Cavanna AE. The pharmacology of Tourette syndrome. J Neural Transm (Vienna). 2013 Apr;120(4):689-94. doi: 10.1007/s00702-013-0979-z. Epub 2013 Jan 30. PMID 23361655
- [Background] Scahill L, Woods DW, Himle MB, Peterson AL, Wilhelm S, Piacentini JC, McNaught K, Walkup JT, Mink JW. Current controversies on the role of behavior therapy in Tourette syndrome. Mov Disord. 2013 Aug;28(9):1179-83. doi: 10.1002/mds.25488. Epub 2013 May 16. PMID 23681719
- [Background] Lin L, Stamm K, Christidis P, APA Center for Workforce Studies. 2015 County-Level Analysis of U.S. Licensed Psychologists and Health Indicators [online]. 2016. Available at: http://www.apa.org/workforce/publications/15-county-analysis/index.aspx?tab=1 Accessed 9/29/2017.
- [Background] Cuenca J, Glazebrook C, Kendall T, Hedderly T, Heyman I, Jackson G, Murphy T, Rickards H, Robertson M, Stern J, Trayner P, Hollis C. Perceptions of treatment for tics among young people with Tourette syndrome and their parents: a mixed methods study. BMC Psychiatry. 2015 Mar 11;15:46. doi: 10.1186/s12888-015-0430-0. PMID 25879205
- [Background] Morera Maiquez B, Sigurdsson HP, Dyke K, Clarke E, McGrath P, Pasche M, Rajendran A, Jackson GM, Jackson SR. Entraining Movement-Related Brain Oscillations to Suppress Tics in Tourette Syndrome. Curr Biol. 2020 Jun 22;30(12):2334-2342.e3. doi: 10.1016/j.cub.2020.04.044. Epub 2020 Jun 4. PMID 32502412
- [Derived] Iverson AM, Arbuckle AL, Song DY, Bihun EC, Black KJ. Median Nerve Stimulation for Treatment of Tics: A 4-Week Open Trial with Ecological Momentary Assessment. J Clin Med. 2023 Mar 28;12(7):2545. doi: 10.3390/jcm12072545. PMID 37048629
- See also: Invitation to participate — https://tics.wustl.edu/participate/median-nerve-stimulation-study/
- Available data/document: Study Protocol: 2y7fs — https://osf.io/2y7fs/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from those 32 participants who completed an in person RCT (randomized controlled trial; registration number NCT04731714). One RCT participant did not choose to participate in this open-label extension. Recruitment occurred between November 2021 and April 2022.
Groups:
- Active MNS: Active, self-directed electrical stimulation of the median nerve: Electrical stimulation of the median nerve (12 Hz, pulse width 200µs), initially at the threshold needed to see movement of the right thumb with right median nerve stimulation. After initial training with the device and education in the rationale for suprathreshold stimulation, participants will choose timing and intensity of stimulation based on their momentary symptom severity and their experience with the treatment since the beginning of the study. Participant can choose right or left median nerve (we will suggest their nondominant hand to minimize interference with daily activities).
Period: Overall Study
Arm/Group | Active MNS
Started | 31
Completed At Least 1 EMA (Ecological Momentary Assessment) Survey | 30
Completed | 27
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Everyone who signed an informed consent document for this study.
Arm/Group | Active MNS
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Time Spent Using the Device Per Day of Use
Description: Number of minutes per day the device was used, only counting days in which the device was turned on, over the four-week period after the initial visit
Time Frame: At study conclusion, up to 4 weeks
Measure: Median (Inter-Quartile Range); unit: minutes per day
Arm/Group | Active MNS
Number analyzed (Participants) | 31
minutes per day | 49.6 [24.2 to 117.2]

2. Primary Outcome: Time Spent Using the Device (Days Per Week)
Description: Number of days per week the device was used
Time Frame: At study conclusion, up to 4 weeks
Population: All participants enrolled in study
Measure: Median (Inter-Quartile Range); unit: days per week
Arm/Group | Active MNS
Number analyzed (Participants) | 31
days per week | 1.5 [0.6 to 2.0]

3. Primary Outcome: Plan to Continue MNS (Median Nerve Stimulation)
Description: Answered yes (from options yes / no / maybe) to the question, "Do you expect to continue to use the stimulator?"
Time Frame: At study conclusion, up to 1 month
Population: All participants who completed the final survey
Measure: Count of Participants; unit: Participants
Arm/Group | Active MNS
Number analyzed (Participants) | 27
Participants | 21

4. Primary Outcome: Change in Tic Frequency With Stimulation
Description: Change in self-reported tic frequency on the frequency item (score range from 0 = no tics [better] to 5 = always [worse]) from the Yale Global Tic Severity Scale (YGTSS) from the beginning to the end of each stimulation period. Participants were instructed to answer this question every time they turned on the device and every time they turned it off, every day for 4 weeks. The difference between the turning off score and the previous turning on score was averaged across all ratings completed during the 4 weeks of the trial. The wording of the score anchors is provided at https://osf.io/7pjk4 .
Time Frame: Recorded every time the device was turned on and every time it was turned off, up to 4 weeks
Population: All participants with at least one on-off survey pair during the study period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active MNS
Number analyzed (Participants) | 25
score on a scale
  All participants "turning ON" surveys | 3.1 (1.0)
  All participants "turning OFF" surveys | 2.1 (1.1)
Statistical Analysis 1: Comparison: Active MNS; Test type: Superiority; p < 0.001, t-test, 2 sided; paired t-test
Statistical Analysis 2: Comparison: Active MNS; Correlation of this Outcome measure (change in tic frequency with stimulation during this study) with the change in tic frequency (measured as the number of 10-second tic-free intervals) during active, rhythmic stimulation in the randomized, controlled trial of MNS that all participants had previously completed; Test type: Other — Pearson correlation test; p = 0.33, Regression, Linear; Pearson's R; Pearson's R = 0.21, 95% CI 2-sided [-0.22 to 0.56]

5. Primary Outcome: Change in Tic Intensity With Stimulation
Description: Change in self-reported tic intensity on the intensity item (score range from 0 = no tics [better] to 5 = severe intensity [worse]) from the Yale Global Tic Severity Scale (YGTSS) from the beginning to the end of each stimulation period. Participants were instructed to answer this question every time they turned on the device and every time they turned it off, every day for 4 weeks. The difference between the turning off score and the previous turning on score was averaged across all ratings completed during the 4 weeks of the trial.
Time Frame: Recorded every time the device was turned on and every time it was turned off, up to 4 weeks
Population: All participants with at least one on-off survey pair during the study period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active MNS
Number analyzed (Participants) | 25
score on a scale
  All participants "turning ON" surveys | 2.9 (0.8)
  All participants "turning OFF" surveys | 2.0 (1.1)
Statistical Analysis 1: Comparison: Active MNS; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Paired Samples Wilcoxon Test
Statistical Analysis 2: Comparison: Active MNS; Correlation of this Outcome measure (change in tic intensity during this study) with change in tic intensity during active, rhythmic stimulation during the randomized, controlled trial that all participants had previously completed; Test type: Other — Pearson's R; p = 0.08, Regression, Linear; Pearson's R; Pearson's R = 0.36, 95% CI 2-sided [-0.05 to 0.66]

6. Primary Outcome: Discomfort
Description: Mean discomfort while using the stimulator, on a 0-3 scale adapted from the Clinical Global Impression - Improvement [CGI-I] Efficacy Index. Specifically, the prompt was "How much DISCOMFORT did the stimulation cause?", and the participant selected one of the following responses:
  0 = NO discomfort
  1. = discomfort noticeable, but not severe enough to concern me or to turn it off
  2. = enough discomfort, impairment of functioning or social embarrassment that I would only keep it on if the benefit was considerable
  3. = caused discomfort, impairment of functioning or social embarrassment to a degree that any treatment benefit was not worth leaving it on Higher values represent a worse outcome. Discomfort was reported at the end of each stimulation period, and at random times twice daily between 9a.m. and 9p.m. when prompted by text message, if the device was on when the text was received.
Time Frame: Recorded every time the device was turned off, and every time the participant was prompted by a text to fill out the survey if the device was on when the text was received, up to 4 weeks.
Population: All participants who completed the discomfort question at least once during the study after initial training.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active MNS
Number analyzed (Participants) | 26
units on a scale | 1.0 [0.6 to 1.5]

7. Secondary Outcome: CGI-I (Clinical Global Impression--Improvement)
Description: Overall impact of the stimulation on symptoms throughout the study period:
  1. = Very much improved - nearly all better; good level of functioning; minimal symptoms; represents a very substantial change
  2. = Much improved - notably better with significant reduction of symptoms; increase in the level of functioning but some symptoms remain
  3. = Minimally improved - slightly better with little or no clinically meaningful reduction of symptoms. Represents very little change in basic clinical status, level of care, or functional capacity
  4. = No change - symptoms remain essentially unchanged
  5. = Minimally worse - slightly worse but may not be clinically meaningful; may represent very little change in basic clinical status, level of care, or functional capacity
  6. = Much worse - clinically significant increase in symptoms and diminished functioning
  7. = Very much worse - severe exacerbation of symptoms and loss of functioning On this scale, lower numbers indicate a better outcome.
Time Frame: At study conclusion, up to 4 weeks
Population: All participants who completed the final survey.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active MNS
Number analyzed (Participants) | 27
units on a scale | 3.1 [2.7 to 3.4]

8. Secondary Outcome: CGI Efficacy Index: Side Effects
Description: Overall discomfort from stimulation throughout the study period. The prompt for this survey question was: "On average, over the course of the study, how much DISCOMFORT did the stimulation cause? (If discomfort is the wrong word, please substitute any negative effects or side effects of stimulation.)" Participants chose one of the following answers:
  0 no discomfort
  1. discomfort noticeable, but not severe enough to concern me or to turn it off
  2. enough discomfort, impairment of functioning or social embarrassment that I would only keep it on if the benefit was considerable
  3. caused discomfort, impairment of functioning or social embarrassment to a degree that any treatment benefit was not worth leaving it on On this scale, lower numbers represent a better outcome.
Time Frame: At study conclusion, up to 4 weeks
Population: All participants who completed the final survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active MNS
Number analyzed (Participants) | 27
units on a scale | 1.2 (1.0)

9. Secondary Outcome: Mean Therapeutic Effect During Stimulator Use
Description: Mean self-rated therapeutic effect (from the modified CGI Efficacy Index) when device is on, reported at the end of the study. Specifically, the prompt for this question was "On average, over the course of the study, how much did your tics IMPROVE during stimulation?" Participants chose one of the following answers:
  0 Unchanged or worse
  1. Minimal - Slight improvement that doesn't decrease the overall impact of symptoms.
  2. Moderate - Decided improvement. Partial remission of symptoms
  3. Marked - Vast improvement. Complete or nearly complete remission of all symptoms On this scale, higher numbers represent a better outcome.
Time Frame: At study conclusion, up to 4 weeks
Population: All participants who completed the final survey.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active MNS
Number analyzed (Participants) | 27
units on a scale | 1.5 [1.1 to 1.9]

10. Secondary Outcome: Change in Self-reported Tic Severity
Description: Self-rated tic severity over the past week using the Adult Tic Questionnaire (ATQ), first rating at (or within 2 weeks prior to) the beginning of study participation and second rating at the end of study participation. Higher ATQ scores reflect a worse outcome. For each tic present in the past week, its severity score is the sum of its frequency score (0-4, 4 worst, occurring "almost all the time during the day") and its intensity score (0-4, 4 worst). The ATQ severity score is the sum of the severity score for each of up to 27 tics present in the past week. The minimum possible severity score on the ATQ is 0, indicating that no tics were present in the past week. The maximum possible severity score on the ATQ indicates is 216, indicating that a tic of each of the 27 types listed was present in the past week, each with an item severity score of 8 = 4 + 4.
Time Frame: At beginning of study participation or up to 2 weeks prior, and again at end of study participation up to 4 weeks
Population: All participants with ATQ scores both at baseline and during final survey (those who completed final survey more than 4 weeks after completing the study were excluded).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active MNS
Number analyzed (Participants) | 25
units on a scale
  baseline score | 35.4 (16.7)
  final survey score | 34.6 (22.5)
Statistical Analysis 1: Comparison: Active MNS; Test type: Other — Traditional comparative; p = 0.84, Paired Sample t-Test, 2-Sided

11. Secondary Outcome: Self-reported Duration of MNS Benefit, in Minutes
Description: On the survey at the end of study participation, the relevant question asked: "On average, over the course of the study, how long do you think the improvement in your tics lasted after you turned off the device? Give answer in minutes. Enter 0 (zero) if improvement with stimulation stopped immediately when you turned the device off." On this item, higher answers indicate a better outcome.
Time Frame: Monitored over the entire period of study participation, up to 4 weeks
Population: All participants who answered this question on the final survey
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Active MNS
Number analyzed (Participants) | 21
minutes | 15 [10 to 45]

ADVERSE EVENTS:
Time Frame: through study completion, up to 4 weeks
Description: Data were collected by open-ended question on the final survey regarding the full period of time up to four weeks from enrollment through completing the final survey.
Arm/Group | Active MNS
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 4/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active MNS (N=31)
Skin Irritation (Skin and subcutaneous tissue disorders) | 2
Stimulation Limited Muscle Dexterity (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT05016765/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT05016765/ICF_000.pdf